CLINICAL TRIAL: NCT06221891
Title: Early Evaluation of Left Ventricular Systolic Function Impairment in Patients With Chronic Kidney Disease by Multimodal Ultrasonography
Status: Recruiting | Type: Observational
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.CSK.006
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Chronic Kidney Diseases; Left Ventricular Systolic Dysfunction
Keywords: first phase ejection fraction;left ventricular systolic dysfunction;echocardiography;chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: This group contains the patients with chronic kidney disease.
- control group: This group contains the healthy adults.

SUMMARY:
The goal of this observational study is to learn about the value of multimodal ultrasound in early detection of left ventricular systolic dysfunction in patients with chronic kidney disease(CKD). The main questions it aims to answer are:

1. If first-phase ejection fraction（EF1）could early detect the left ventricular systolic dysfunction in patients with CKD.
2. Whether EF1 can detect left ventricular systolic dysfunction in patients with CKD more sensitively than speckle-tracking echocardiography and myocardial work.

Participants will need to cooperate to do an echocardiography. Researchers will compare healthy volunteers and patients with CKD to see if EF1 could early detect the left ventricular systolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease who are hospitalized in The Fifth Affiliated Hospital of Sun Yat-sen University.
* LVEF≥50%.

Exclusion Criteria:

* Patients with primary hypertension, diabetes and congenital heart disease.
* Patients who are pregnant or lactating.
* Patients with the blurry ultrasound images.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who are hospitalized in The Fifth Affiliated Hospital of Sun Yat-sen University.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
first-phase ejection fraction | 1 hour
  an ultrasound indicator used to assess early left ventricular systolic function

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China